CLINICAL TRIAL: NCT05028205
Title: Eating Better Together: A Pilot Study
Brief Title: EBT Fruit and Vegetable Prescription
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Tennessee, Knoxville (Other)
Responsible Party: Principal Investigator, Hollie Raynor, Associate Dean of Research for the College of Education, Health, and Human Sciences, The University of Tennessee, Knoxville
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UTK IRB-21-06251-FB
Record Dates: First submitted 2021-08-16; First posted 2021-08-31 (Actual); Last update posted 2025-04-03 (Actual); Status verified 2025-04

CONDITIONS: Childhood Obesity; Obesity
Keywords: Fruit and Vegetable Prescription; Food Security
MeSH Terms: conditions — Pediatric Obesity; Obesity

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Prevention Plus (Experimental): Child's energy balance behavioral goals will be to consume < 3 sugar-sweetened beverages (e.g., regular carbonated soft drinks, sports drinks, lemonades, ice teas, flavored milk, juice drinks < 100% juice, and punches) servings /wk, ≥1 1/2 cups/day of whole vegetables and ≥ 1 cup/day of whole fruit, engage in ≥ 60 minutes/day of moderate- to vigorous-intensity physical activity, and reduce TV viewing to < 2 hours/day. The caregiver's energy balance behavioral goals will be to consume < 3 sugar-sweetened beverage servings/wk, ≥ 2 1/2 cups/day of whole vegetables and ≥ 1 1/2 cups/day of whole fruit, engage in ≥ 150 minutes of moderate- to vigorous-intensity physical activity per week and reduce TV viewing to < 10 hours/wk.
  Interventions: Behavioral: Prevention Plus

INTERVENTIONS:
Behavioral: Prevention Plus — Families will receive a behavioral intervention for childhood obesity provided by a BHC. This will consist of three, in-person meetings (months 1, 3, and 5), and three, 20-minute phone calls (months 2,4, and 6). During in-person visits, child height and weight will be taken, and BMI will be plotted on the BMI-for-age growth chart. During these sessions, families will receive feedback on child growth and weight status. Prevention Plus materials and child and caregiver energy balance behavior goals will be reviewed. The phone calls will be with the caregiver, where caregivers will be asked to measure the height and weight of their child, calculate BMI, and plot on the BMI-for-age growth chart. The BHC will discuss the family's progress on achieving child and caregiver goals and implementation of behavioral parenting strategies. Families will receive a fruit and vegetable prescription (FVx) in addition to the standard Prevention Plus family-based behavioral weight loss treatment.

SUMMARY:
Eating Better Together is a 6-month pilot program that teaches families about healthy eating and activity and provides home deliveries of fresh fruits and vegetables from a local retail partner.

DETAILED DESCRIPTION:
Efficacious primary care-based childhood overweight/obesity interventions for children from low-income homes are needed to address health disparities. The University of Tennessee (UT) and Cherokee Health Systems (CHS), a federally qualified health center, has piloted a 6-month childhood overweight/obesity intervention for underserved children (R34DK109504). The intervention was based upon Prevention Plus, the recommended primary care-based treatment for childhood overweight/obesity, which includes targeting fruit and vegetable (FV) and sugar-sweetened beverage intake, physical activity, and screen time; incorporates behavior modification techniques, and uses a family-based approach. The intervention structure was designed to reduce family costs related to time, thus monthly contact alternated between in-person sessions and phone calls, and in-person sessions could occur using "warm hand-offs" between providers (allowed piggybacking of appointments). The pilot demonstrated CHS' ability to implement the intervention using their electronic health record (EHR). The intervention significantly reduced child standardized BMI (ZBMI).

While the intervention reduced ZBMI, the degree of reduction was below what is recommended to achieve cardiometabolic improvements in children (-0.25 ZBMI). Families (58.9% with a household income of < $20,000/yr, 32.9% with household food insecurity, 50.7% receiving SNAP benefits, and 94.5% receiving free or reduced-price school meals) reported problems with having enough food, particularly FVs, which was a barrier for intervention participation. Thus, increasing the affordability of FVs may enhance the achievement of intervention dietary goals, which should increase diet quality and enhance ZBMI reduction.

One method to increase FV affordability is a prescription incentive program. In these programs, a "prescription," often for FVs, from a health care provider is given to the participant, and the prescription includes delivery of fresh FVs to the family's home. Adult FV prescription studies have reported increases in FV intake and decreases in BMI. In children, three uncontrolled studies reported that an FV prescription program increased FV intake, with the influence on child weight status not reported. Thus, to enhance the efficacy of our 6-month Prevention Plus intervention in addressing health disparities in childhood overweight/obesity, investigators will pilot test Prevention Plus, our tested intervention, with the addition of an FV prescription incentive program (Prevention Plus+FVx). For Prevention Plus+FVx, to assist families in achieving FV goals (FV prescription), they will receive up to $60/month ($1/day for each child and parent) deliveries of fresh FVs to their home from a local retail partner (Food City). Thirty families receiving their primary care from CHS, with an adult caregiver and a child aged 4 to 10 years with a BMI > 85th percentile, will participate in the program.

Participants

CHS families eligible for the trial will be patients at the CHS Knox County Pediatric Clinic. Additional eligibility criteria include families with a child who is aged 4 to 10 years, with a BMI > 85 percentile, who have an adult (> 18 years) caregiver living in the household willing to participate in the program. The adult caregiver needs to be able to read and speak English; and be willing to shop for fresh fruits and vegetables at the Western Ave Food City store (1950 Western Ave., Knoxville, TN, 37921).

Recruitment

For recruitment, the EHR, via the client dashboard, will alert if a family is eligible when the EHR is opened by any primary care provider. This alert will prompt the provider to conduct a "warm hand-off" of the family to the Behavioral Health Consultant (BHC) in the clinic to start the enrollment process. The BHC will discuss the study with the family and will ask interested families to write their name and phone number at the bottom of an eligibility form, which will indicate that the family would like to be contacted by the research team. BHCs will provide families with a flyer about the program. After BHCs discuss the program with families, they will complete a template in the EHR indicating the enrollment status of the family. This will allow the EHR to give an appropriate alert (or not) to physicians in the future about the need (or not) of the "warm hand-off" of the family to the BHC.

Research staff will engage with interested potential participants in two ways. The first option is an in-person greeting at Cherokee Mills, an office campus that houses both the CHS Knox County Pediatric Clinic and a UT office space. When research staff are present at UT's Cherokee Mills office, BHCs will be able to introduce interested families to research staff in-person. If the family is interested and available, research staff can provide a study overview, complete an eligibility screening, and schedule an orientation session at that time. When staff are not present at Cherokee Mills, completed eligibility forms will be sent to the lead BHC at CHS, who will securely send scanned copies of the documents to Dr. Raynor's research team using Vault, UT's secure file transmission service. Once scanned/sent the original copies will be destroyed/shredded by the lead BHC at CHS. Interested potential families will be contacted by the research team and phone screened for eligibility. Eligible families will be invited to an orientation.

Orientations will be at in-person at UT's campus or UT's office space at Cherokee Mills, or online via Zoom, depending on the family's preference. All in-person meetings will follow any health safety procedures that are in place at the time of the meeting. The orientations sessions will occur one-on-one between a family and a research team member. Families will be mailed/emailed the consent forms prior to the orientation. For potential families who are interested, the research team will review the consent form at the end of the orientation and adult caregivers will sign consent forms and children will provide assent (verbal or written). Families that are engaging in the orientation online via Zoom will sign the consent/assent form on Qualtrics.

Baseline Assessment

Following the signing of the consent form, the complete baseline assessment will occur. This will include the completion of all questionnaires and measures of anthropometrics.

For orientations occurring online, following the signing of the consent form, questionnaires will be completed by verbally reviewing the questionnaires with families and collecting responses. An appointment will be set-up to collect height and weight (anthropometrics) measures at the participant's home or at UT's campus or the UT's office space at Cherokee Mills (the location will depend on participant preference). These meetings will follow health safety procedures in place at the time.

Study/Project Procedures

Following baseline assessment, families will begin the intervention. Children will continue to receive standard care at CHS. After attendance to the first intervention session (the 30-minute session in month 1 delivered by the BHC), families will receive a monthly newsletter on general nutrition topics (such as MyPlate or the Dietary Guidelines for Americans). Additionally, each family will receive a scale; a BMI-for-age growth chart; a binder for intervention materials; a self-monitoring diary to record the child's monthly height, weight, BMI, and BMI percentile; and picture-based diaries to monitor daily energy balance behaviors. Additional family materials will be included in the EHR template for each session. Family materials provided at each session will outline a process to measure growth and include information about how children grow, as well as cover behavioral parenting strategies to assist with changing child behavior (self-monitoring, modeling [caretakers will be asked to make and monitor the same energy balance behavior changes as their child], stimulus control, and positive reinforcement) for energy balance behaviors. These behavioral parenting strategies are based upon Social Cognitive Theory. Sessions will be written at the fifth-grade reading level.

Families will meet in person or via telehealth appointment (depending on the current standard of care at CHS, and University of Tennessee policy-- meaning that when CHS or UT has a policy place that does not allow in-person contact, investigators will hold these appointments via telehealth, when these policies are not in effect, the family can choose to attend the appointment in-person or via telehealth) with a BHC at the CHS clinic in which they receive care for 30 minutes during months 1, 3, and 5. In these sessions, child height and weight will be taken, and BMI will be plotted on the BMI-for-age growth chart. Families will receive feedback about growth and the weight status of their child. Additionally, the session materials will be reviewed and behavioral parenting strategies will be encouraged to aid with changing two dietaryy and two leisure-time activity (energy balance) behaviors of the child. As is traditional in a family-based approach, the caregiver will also change the same energy balance behaviors as the child, as adult caregivers can then model healthy behaviors for the child, assisting the child in learning the new weight-related behaviors. Thus, both the caregiver and child will be encouraged to change and self-monitor energy balance behaviors with the use of the picture-based diaries. Achievement of energy balance behavior goals of both the child and the caregiver will be reviewed (via the picture-based diaries) and BHCs will problem-solve areas to assist families with achieving goals, suggesting the use of the behavioral parenting strategies as needed.

During months 2, 4, and 6, BHCs will complete a 20-minute phone call with the caregiver. Caregivers will be asked to measure the height and weight of their child, calculate BMI and plot it on the BMI-for-age growth chart prior to the call. During the call, the BHC will provide feedback on the changes in child growth since the previous contact. Additionally, the BHC will discuss the family's progress on achieving child and caregiver energy balance behavior goals and implementation of behavioral parenting strategies.

The child's energy balance behavioral goals will be to consume < 3 sugar-sweetened beverages (e.g., regular carbonated soft drinks, sports drinks, lemonades, ice teas, flavored milk, juice drinks < 100% juice, and punches) servings /wk, ≥1 1/2 cups/day of whole vegetables and ≥ 1 cup/day of whole fruit, engage in ≥ 60 minutes/day of moderate- to vigorous-intensity physical activity, and reduce TV viewing to < 2 hours/day. The caregiver's energy balance behavioral goals will be to consume < 3 sugar-sweetened beverage servings/wk, ≥ 2 1/2 cups/day of whole vegetables and ≥ 1 1/2 cups/day of whole fruit, engage in ≥ 150 minutes of moderate- to vigorous-intensity physical activity per week and reduce TV viewing to < 10 hours/wk. To increase self-efficacy, the goals will be incrementally increased, with families implementing the full program goals at month four. Additionally, children and caregivers will be asked to achieve at least three of the five goals each day (child) or week (adult caregiver). The cost will be considered in all sessions, with BHC's providing low-cost options for achieving goals (purchasing canned or frozen fruits and vegetables to eat instead of fresh fruits and vegetables).

To help children and families meet their goals-particularly their dietary goals related to fruit and vegetable consumption-- families will receive a fruit and vegetable prescription (FVx) in addition to the standard Prevention Plus family-based behavioral weight loss treatment. The FVx will include home deliveries of fresh FVs from our retail grocery partner (Food City), up to $60/month for each session attended. Families will have access to the $60 for one month and then it will expire. Families will receive weekly texts that include available delivery windows, remaining funds for the month, and reminders of expiration date.

ELIGIBILITY:
Inclusion Criteria:

* Patients at the Cherokee Health Systems clinic in Cherokee Mills
* Child age between 4 to 10 years old
* Child BMI > 85th percentile
* Child must have an adult caregiver (> 18 years) living in the household and be willing to participate in the program
* Adult caregivers need to be able to read and speak English

Exclusion Criteria:

* Not patients at the CHS Knox County Pediatric Clinic
* A child not within the 4 to 10 years age range
* Child BMI at or below the 85 percentile
* Child without an adult caregiver (> 18 years) living in the household and not willing to participate in the program
* Adult caregivers that are not able to read and speak English

Ages: 4 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 30 (Estimated)
Dates: Start 2021-08-16 (Actual); Primary Completion 2026-02-02 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Project Reach, the number of participants who participate in the study | through study completion, an average of 6 months
  Measurement in project reach will aid in the evaluation of the implementation process for the study, and will help us determine the feasibility of a larger study. Reach will be determined using the data from the EHR at CHS. Specifically, investigators will use data reports from the EHR to determine the number of participants who participate in the study.
Project Reach, participants who are eligible to participate in this study, but decline to participate in the study | through study completion, an average of 6 months
  Measurement in project reach will aid in the evaluation of the implementation process for the study, and will help us determine the feasibility of a larger study. Reach will be determined using the data from the EHR at CHS. Specifically, investigators will use data reports from the EHR to determine the number of participants who are eligible to participate in this study, but decline to participate in the study.
Project Reach, total number of participants/patients who meet eligibility criteria | through study completion, an average of 6 months
  Measurement in project reach will aid in the evaluation of the implementation process for the study, and will help us determine the feasibility of a larger study. Reach will be determined using the data from the EHR at CHS. Specifically, investigators will use data reports from the EHR to determine the total number of participants/patients who meet the eligibility criteria for the study.
Intervention Session Completion | through study completion, an average of 6 months
  Completion of the number of each intervention session will be documented in the EHR.
Funds spent on FV deliveries | through study completion, an average of 6 months
  Looking at total amount spent of FV deliveries will help us to identify if the fruit and vegetable prescription program was implemented as intended.

SECONDARY OUTCOMES:
Demographics | Baseline only
  Will be assessed and used to describe the study sample. Demographics collected will include: child and caregiver measures of age, gender, race/ethnicity, and caregiver measures of marital status, caregiver education level, employment status, and income.
Household Information | Change from baseline and through study completion, an average of 6 months
  The number of people living in the household and federal food program participation (e.g., SNAP, WIC, NSLP) will be collected.
Food Purchasing and Household Food Availability | Change from baseline and through study completion, an average of 6 months
  This assessment asks participants about food purchasing habits and to report of selected common food and beverage items had been purchased for the household in the last month, as well as, if the food or beverage item is available in the home. This assessment will allow us to explore differences in food purchasing patterns, and differences in the healthfulness of the food/beverages available in the home before and after the provision of the weight management intervention with fruit and vegetable home deliveries.
Food Security | Change from baseline and through study completion, an average of 6 months
  Food security will be assessed using the gold-standard, USDA food security modules to test for food insecurity in both adults and children in a household.
Dietary Intake of Fruits and Vegetables | Change from baseline and through study completion, an average of 6 months
  The National Cancer Institute's fruit and vegetable dietary screener will be administered to child participants to determine if there are changes in dietary intake of fruits and vegetables. The screener will be completed by the child participant and by the adult caregiver.
Beverage Intake | Change from baseline and through study completion, an average of 6 months
  Child beverage intake in the last month will be assessed via the BEV-Q. This will be completed for the child participant and the adult caregiver.
Anthropometrics | Change from baseline and through study completion, an average of 6 months
  Child and adult caregiver heights and weights will be measured to calculate BMI and asses changes in BMI z-scores.

CONTACTS AND LOCATIONS:
Overall Officials: Hollie A Raynor, PhD, Principal Investigator — University of Tennessee, Knoxville
Locations (2):
- United States (2):
  - Cherokee Health Systems, Dameron Avenue Pedatrics, Knoxville, Tennessee
  - Healthy Eating and Activity Laboratory, Knoxville, Tennessee

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Skinner AC, Ravanbakht SN, Skelton JA, Perrin EM, Armstrong SC. Prevalence of Obesity and Severe Obesity in US Children, 1999-2016. Pediatrics. 2018;141(3):e20173459. Pediatrics. 2018 Sep;142(3):e20181916. doi: 10.1542/peds.2018-1916. No abstract available. PMID 30177517
- [Background] Ogden CL, Carroll MD, Fakhouri TH, Hales CM, Fryar CD, Li X, Freedman DS. Prevalence of Obesity Among Youths by Household Income and Education Level of Head of Household - United States 2011-2014. MMWR Morb Mortal Wkly Rep. 2018 Feb 16;67(6):186-189. doi: 10.15585/mmwr.mm6706a3. PMID 29447142
- [Background] Whitaker RC, Pepe MS, Wright JA, Seidel KD, Dietz WH. Early adiposity rebound and the risk of adult obesity. Pediatrics. 1998 Mar;101(3):E5. doi: 10.1542/peds.101.3.e5. PMID 9481024
- [Background] Whitaker RC, Wright JA, Pepe MS, Seidel KD, Dietz WH. Predicting obesity in young adulthood from childhood and parental obesity. N Engl J Med. 1997 Sep 25;337(13):869-73. doi: 10.1056/NEJM199709253371301. PMID 9302300
- [Background] Demmer RT, Zuk AM, Rosenbaum M, Desvarieux M. Prevalence of diagnosed and undiagnosed type 2 diabetes mellitus among US adolescents: results from the continuous NHANES, 1999-2010. Am J Epidemiol. 2013 Oct 1;178(7):1106-13. doi: 10.1093/aje/kwt088. Epub 2013 Jul 25. PMID 23887044
- [Background] Menke A, Casagrande S, Geiss L, Cowie CC. Prevalence of and Trends in Diabetes Among Adults in the United States, 1988-2012. JAMA. 2015 Sep 8;314(10):1021-9. doi: 10.1001/jama.2015.10029. PMID 26348752
- [Background] Seburg EM, Olson-Bullis BA, Bredeson DM, Hayes MG, Sherwood NE. A Review of Primary Care-Based Childhood Obesity Prevention and Treatment Interventions. Curr Obes Rep. 2015 Jun;4(2):157-73. doi: 10.1007/s13679-015-0160-0. PMID 26213643
- [Background] Barlow SE, Dietz WH. Obesity evaluation and treatment: Expert Committee recommendations. The Maternal and Child Health Bureau, Health Resources and Services Administration and the Department of Health and Human Services. Pediatrics. 1998 Sep;102(3):E29. doi: 10.1542/peds.102.3.e29. PMID 9724677
- [Background] Spear BA, Barlow SE, Ervin C, Ludwig DS, Saelens BE, Schetzina KE, Taveras EM. Recommendations for treatment of child and adolescent overweight and obesity. Pediatrics. 2007 Dec;120 Suppl 4:S254-88. doi: 10.1542/peds.2007-2329F. PMID 18055654
- [Background] Dougherty D, Conway PH. The "3T's" road map to transform US health care: the "how" of high-quality care. JAMA. 2008 May 21;299(19):2319-21. doi: 10.1001/jama.299.19.2319. No abstract available. PMID 18492974
- [Background] Raynor HA, Osterholt KM, Hart CN, Jelalian E, Vivier P, Wing RR. Efficacy of U.S. paediatric obesity primary care guidelines: two randomized trials. Pediatr Obes. 2012 Feb;7(1):28-38. doi: 10.1111/j.2047-6310.2011.00005.x. Epub 2011 Dec 13. PMID 22434737
- [Background] Looney SM, Raynor HA. Examining the effect of three low-intensity pediatric obesity interventions: a pilot randomized controlled trial. Clin Pediatr (Phila). 2014 Dec;53(14):1367-74. doi: 10.1177/0009922814541803. Epub 2014 Jul 7. PMID 25006118
- [Background] Altman M, Wilfley DE. Evidence update on the treatment of overweight and obesity in children and adolescents. J Clin Child Adolesc Psychol. 2015;44(4):521-37. doi: 10.1080/15374416.2014.963854. Epub 2014 Dec 12. PMID 25496471
- [Background] US Preventive Services Task Force; Grossman DC, Bibbins-Domingo K, Curry SJ, Barry MJ, Davidson KW, Doubeni CA, Epling JW Jr, Kemper AR, Krist AH, Kurth AE, Landefeld CS, Mangione CM, Phipps MG, Silverstein M, Simon MA, Tseng CW. Screening for Obesity in Children and Adolescents: US Preventive Services Task Force Recommendation Statement. JAMA. 2017 Jun 20;317(23):2417-2426. doi: 10.1001/jama.2017.6803. PMID 28632874
- [Background] Guideline Development Panel for Treatment of Obesity, American Psychological Association. Summary of the clinical practice guideline for multicomponent behavioral treatment of obesity and overweight in children and adolescents. Am Psychol. 2020 Feb-Mar;75(2):178-188. doi: 10.1037/amp0000530. PMID 32052993
- [Background] Krebs-Smith SM, Pannucci TE, Subar AF, Kirkpatrick SI, Lerman JL, Tooze JA, Wilson MM, Reedy J. Update of the Healthy Eating Index: HEI-2015. J Acad Nutr Diet. 2018 Sep;118(9):1591-1602. doi: 10.1016/j.jand.2018.05.021. PMID 30146071
- [Background] Perry CP, Keane E, Layte R, Fitzgerald AP, Perry IJ, Harrington JM. The use of a dietary quality score as a predictor of childhood overweight and obesity. BMC Public Health. 2015 Jun 24;15:581. doi: 10.1186/s12889-015-1907-y. PMID 26100985
- [Background] Thomas JG, Doshi S, Crosby RD, Lowe MR. Ecological momentary assessment of obesogenic eating behavior: combining person-specific and environmental predictors. Obesity (Silver Spring). 2011 Aug;19(8):1574-9. doi: 10.1038/oby.2010.335. Epub 2011 Jan 27. PMID 21273995
- [Background] Thomas JG, Bond DS, Raynor HA, Papandonatos GD, Wing RR. Comparison of Smartphone-Based Behavioral Obesity Treatment With Gold Standard Group Treatment and Control: A Randomized Trial. Obesity (Silver Spring). 2019 Apr;27(4):572-580. doi: 10.1002/oby.22410. Epub 2019 Feb 19. PMID 30779333
- [Background] Banks GG, Berlin KS, Rybak TM, Kamody RC, Cohen R. Disentangling the Longitudinal Relations of Race, Sex, and Socioeconomic Status, for Childhood Body Mass Index Trajectories. J Pediatr Psychol. 2016 May;41(4):453-61. doi: 10.1093/jpepsy/jsv062. Epub 2015 Jun 27. PMID 26117140
- [Background] Buscemi J, Murphy JG, Berlin KS, Raynor HA. A behavioral economic analysis of changes in food-related and food-free reinforcement during weight loss treatment. J Consult Clin Psychol. 2014 Aug;82(4):659-69. doi: 10.1037/a0036376. Epub 2014 Mar 24. PMID 24660672
- [Background] Skelton JA, Buehler C, Irby MB, Grzywacz JG. Where are family theories in family-based obesity treatment?: conceptualizing the study of families in pediatric weight management. Int J Obes (Lond). 2012 Jul;36(7):891-900. doi: 10.1038/ijo.2012.56. Epub 2012 Apr 24. PMID 22531090
- [Background] Russ SA, Larson K, Franke TM, Halfon N. Associations between media use and health in US children. Acad Pediatr. 2009 Sep-Oct;9(5):300-6. doi: 10.1016/j.acap.2009.04.006. Epub 2009 Jul 9. PMID 19592321
- [Background] Fulkerson JA, Nelson MC, Lytle L, Moe S, Heitzler C, Pasch KE. The validation of a home food inventory. Int J Behav Nutr Phys Act. 2008 Nov 4;5:55. doi: 10.1186/1479-5868-5-55. PMID 18983668
- [Background] Polacsek M, Moran A, Thorndike AN, Boulos R, Franckle RL, Greene JC, Blue DJ, Block JP, Rimm EB. A Supermarket Double-Dollar Incentive Program Increases Purchases of Fresh Fruits and Vegetables Among Low-Income Families With Children: The Healthy Double Study. J Nutr Educ Behav. 2018 Mar;50(3):217-228.e1. doi: 10.1016/j.jneb.2017.09.013. Epub 2017 Nov 7. PMID 29126661
- [Background] Marcinkevage J, Auvinen A, Nambuthiri S. Washington State's Fruit and Vegetable Prescription Program: Improving Affordability of Healthy Foods for Low-Income Patients. Prev Chronic Dis. 2019 Jul 18;16:E91. doi: 10.5888/pcd16.180617. PMID 31322108
- [Background] Bryce R, Guajardo C, Ilarraza D, Milgrom N, Pike D, Savoie K, Valbuena F, Miller-Matero LR. Participation in a farmers' market fruit and vegetable prescription program at a federally qualified health center improves hemoglobin A1C in low income uncontrolled diabetics. Prev Med Rep. 2017 Jun 27;7:176-179. doi: 10.1016/j.pmedr.2017.06.006. eCollection 2017 Sep. PMID 28702315
- [Background] Buyuktuncer Z, Kearney M, Ryan CL, Thurston M, Ellahi B. Fruit and vegetables on prescription: a brief intervention in primary care. J Hum Nutr Diet. 2014 Apr;27 Suppl 2:186-93. doi: 10.1111/jhn.12109. Epub 2013 May 7. PMID 23651065

DOCUMENTS (1):
  • Informed Consent Form (2023-12-07): https://cdn.clinicaltrials.gov/large-docs/05/NCT05028205/ICF_007.pdf